CLINICAL TRIAL: NCT00613600
Title: Safety and Efficacy of Glucomannan for Weight Loss
Brief Title: Safety and Effectiveness Study of a Fiber Supplement for Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Joyce K Keithley, Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTF-GM
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Overweight; Obesity
Keywords: Safety; Efficacy; Glucomannan; Dietary fiber; Weight loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — (1-6)-alpha-glucomannan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Two 665 mg capsules of glucomannan three times a day for eight weeks
  Interventions: Dietary Supplement: Glucomannan
- 2 (Placebo Comparator): Two capsules of inert microcrystalline cellulose three times a day for eight weeks
  Interventions: Dietary Supplement: Inert microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: Glucomannan — Two 665 mg capsules of glucomannan three times a day for 8 weeks
  Arms: 1
Dietary Supplement: Inert microcrystalline cellulose — Two capsules of inert microcrystalline cellulose three times a day for eight weeks
  Arms: 2

SUMMARY:
Overweight and obesity are serious and growing problems within the United States. The usual approaches to weight loss-dieting, exercise, and behavioral interventions-rarely result in long-term weight loss. Therefore, we will evaluate the safety and efficacy of glucomannan, a fiber supplement that has promising weight loss effects.

DETAILED DESCRIPTION:
The primary objective of this exploratory project is to evaluate the safety and efficacy of a highly viscous, water-soluble fiber supplement, glucomannan, for achieving weight loss in overweight and moderately obese individuals. Overweight and obesity are major public health problems in the U.S. that account for substantial morbidity, mortality, and healthcare costs. Conventional approaches to weight loss are largely ineffective, particularly for long-term weight loss and maintenance. Thus, there is a critical need for safe and effective adjunctive treatments. A few, limited studies suggest that glucomannan supplementation is associated with weight loss, is well-tolerated, and has a favorable safety profile.

In this preliminary study, the target population will be overweight and moderately obese individuals, a population that accounts for nearly 50% of all U.S. adults. The specific aims of the project are to: 1) describe the safety of glucomannan for achieving weight loss in overweight and moderately obese individuals, and 2) describe the efficacy of glucomannan for achieving weight loss in overweight and moderately obese individuals. Participants will take glucomannan supplements daily for eight weeks in a double-blind, placebo-controlled, randomized clinical trial. Safety and efficacy outcome measures include: gastrointestinal symptoms/tolerance, hepatic panel, serum creatinine, weight, body composition, diet intake, hunger/fullness, lipid profile, blood glucose, and C-reactive protein. Examination of the safety and efficacy of glucomannan for achieving weight loss will extend our understanding of additional treatments that may be effective in combating a significant public health problem.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 18 and < or = 65 years
* body mass index (BMI) > or = 25 and < or = 35 at study entry
* speak and understand English (since translated versions of study tools have not been validated)
* for females only: without childbearing potential or negative HCG hormone blood test and use of an appropriate form of contraception
* signed informed consent form and HIPAA research authorization

Exclusion Criteria:

* current use of fiber supplements or intolerance to fiber supplements
* untreated/unstable metabolic conditions known to influence weight status (e.g., hypothyroidism, type 2 diabetes mellitus)
* gastrointestinal disorders that might cause complications or influence motility or satiety (e.g., diverticulitis, inflammatory bowel disease, irritable bowel syndrome, intestinal narrowing or obstruction, difficulty swallowing)
* Stage II hypertension (> or = 160/100 mg Hg) or dyslipidemia (fasting LDL cholesterol > or = 160 mg/dL; total cholesterol > or = 240 mg/dL; triglycerides > 200 mg/dL; HDL < or = 40 mg/dL)
* fasting serum glucose > 126 mg/dL
* acute or unstable cardiovascular, pulmonary, hepatic, renal, or psychiatric disorders
* conditions for which weight loss may not be appropriate (e.g., HIV/AIDS, cancer)
* use of medications that might affect weight or food absorption (e.g., diuretics, glucocorticoids, anorexigenic agents, Orlistat, laxatives)
* use of CAM therapies that might affect weight (e.g., acupuncture, Hoodia)
* weight change of > 5% body weight within 3 months of entry into the study
* active eating disorders or active participation in a weight loss program
* renal function impairment as evidenced by a history of renal disease or a serum creatinine > 2.0 mg/dL
* liver function impairment as evidenced by a history of liver disease or liver enzyme elevations > three times the upper limit of normal (i.e., ALT > 150 u/L and/or AST > 165 u/L)
* evidence of depression as determined by a weighted score of > or = 16 on the Center for Epidemiological Studies Depression Scale (CES-D), as this may affect eating behavior and adherence to the study protocol
* currently consumes > or = 10 alcoholic drinks/week, as determined by self-report
* currently smokes cigarettes due to the effects of nicotine on appetite and C-reactive protein levels
* use of illicit drugs currently or in the last six months, as determined by self-report
* for females only: pregnant, less than 6 months postpartum or 6 months post-termination of pregnancy, or currently lactating, due to lack of safety data in this population

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Weight loss | 8 weeks

SECONDARY OUTCOMES:
Body composition | 8 weeks
Dietary intake | 8 weeks
Hunger and fullness | 8 weeks
Lipid profile | 8 weeks
Fasting blood glucose | 8 weeks
C-reactive protein | 8 weeks
Gastrointestinal symptoms and tolerance | 8 weeks
Hepatic panel | 8 weeks
Serum creatinine | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joyce K Keithley, DNSc, RN, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Keithley JK, Swanson B, Mikolaitis SL, DeMeo M, Zeller JM, Fogg L, Adamji J. Safety and efficacy of glucomannan for weight loss in overweight and moderately obese adults. J Obes. 2013;2013:610908. doi: 10.1155/2013/610908. Epub 2013 Dec 30. PMID 24490058